CLINICAL TRIAL: NCT00424671
Title: An Open-Label Study in Healthy Subjects and in Subjects With Stable Impaired Hepatic Function to Assess the Effect of Moderate Hepatic Impairment on Licarbazepine Pharmacokinetics and Metabolism After a Single Dose of 1000 mg Licarbazepine IR Tablets
Brief Title: Effect of Moderate Hepatic Impairment on the Pharmacokinetics and Metabolism of a Single Dose of Licarbazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIC477D2310
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
MeSH Terms: interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

INTERVENTIONS:
Drug: Licarbazepine

SUMMARY:
This study will assess the influence of moderate hepatic impairment on the pharmacokinetics of licarbazepine after single oral administration in healthy subjects and in subjects with stable impaired hepatic function.

ELIGIBILITY:
Inclusion Criteria:

Control group and hepatically impaired groups:

* Male and/or female subjects between 18 and 65 years of age. Female subjects must be surgically sterilized or postmenopausal (Postmenopausal women must have no regular menstrual bleeding for at least 2 years prior to inclusion. Menopause will be confirmed by a plasma FSH level of >40 IU/L. Female subjects must have been surgically sterilized at least 6 months prior to screening. Surgical sterilization procedures must be supported with clinical documentation made available to sponsor and noted in the Relevant Medical History / Current Medical Conditions section of the CRF)
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. The subjects must be able to provide written informed consent prior to study participation, thus excluding subjects with encephalopathy grade 3 or 4.
* Body mass index (BMI) must be within the range of 18 to 32. For instructions and tables see Appendix 5.

Hepatically impaired group:

* Subjects must have liver cirrhosis (hepatic fibrosis with evidence of either micro- or macro-nodular regeneration) confirmed by imaging techniques, ultrasound, MRI or CT.
* Subjects must have physical signs consistent with a clinical diagnosis of liver cirrhosis (e.g., liver firmness to palpation, splenic enlargement, spider angiomata, palmar erythema, parotid hypertrophy, testicular atrophy, gynecomastia).
* Subjects must have a Child-Pugh Clinical Assessment Score between 7 and 9 at both screening and baseline.
* Vital signs (after 3 minutes resting in a supine position) which are within the following ranges: oral body temperature between 35.0-37.5 °C systolic blood pressure, 100-180 mm Hg diastolic blood pressure, 60-115 mm Hg pulse rate, 60 - 100 bpm
* Subjects with creatinine clearance greater than 50 mL/min (based on Cockcroft and Gault formula)

Control group:

* Subjects must be in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Subjects should be matched to the hepatically impaired group in gender, age (±10%), smoking status, BMI (±10%).
* At Screening, and Baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed after the subject has rested for at least three (3) minutes, and again when required after three (3) minutes in the standing position. Vital signs should be within the following ranges: oral body temperature between 35.0-37.5 °C systolic blood pressure, 90-140 mm Hg diastolic blood pressure, 50-90 mm Hg pulse rate, 40 - 90 bpm When blood pressure and pulse will be taken again after 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic or 10 mm Hg drop in diastolic blood pressure and increase in heart rate (>20 bpm) associated with clinical manifestation of postural hypotension. All blood pressure measurements at other time-points should be assessed with the subject supine, unless stated otherwise in the protocol design, and utilizing the same arm for each determination.

Exclusion Criteria:

Control group and hepatically impaired group:

* Participation in any clinical investigation with experimental drug therapy within four weeks prior to dosing or longer as required by local regulation.
* Donation or loss of 400 mL or more of blood within two months prior to dosing.
* Significant acute, new onset illness (ie, flu, gastroenteritis) within two weeks prior to dosi4. A past medical history or clinically significant ECG abnormalities or a family history (grandparents, parents and siblings) of a prolonged QT-interval syndrome.
* History of hyponatremia or seizures.
* History of autonomic dysfunction.
* Subjects with a consistent, abnormally low total lymphocyte count (< 10% of total white blood cell counts)
* A known hypersensitivity to the drug.
* History of immunocompromise, including a positive HIV (ELISA and Western blot) test result.
* Evidence of active alcohol or drug abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Smokers who report cigarette use of more than 20 cigarettes per day. Urine cotinine levels will be measured during screening.

Hepatically impaired group:

* Subjects with a history of unstable, severe, or clinically significant cardiovascular disease
* Polymorphonuclears <1000/µL or platelets <100'000/µL at inclusion.
* Subjects with clinically significant abnormal findings, not consistent with underlying disease, upon physical examination, ECG or laboratory evaluation.
* Subjects with frank symptoms of encephalopathy or ataxia.
* A recent history of acute or chronic bronchospastic disease, including asthma and chronic obstructive pulmonary disease, treated or not treated.
* Any surgical or medical condition which might significantly alter the absorption, distribution, or excretion of any drug.
* Current drug treatment with other mood stabilizers, psychotropic drugs and antiepileptics.

Patients must be willing and able to forgo treatment with restricted medications throughout the study. Approved prescription medications will be allowed during the course of the study on a case by case basis only if the patient has been on a standard treatment regimen for at least 3 months and will continue their regular regimen without change throughout the study (unless required by protocol or to treat an adverse event) Treatments in table 5.1 are allowed in the hepatically impaired group only.

Control group

* Use of any prescription medication within 1 month prior to dosing.
* Use of over-the-counter medications or vitamins during 14 days prior to dosing (Paracetamol, aspirin or ibuprofen are acceptable, but must be documented in the CRF).
* History or presence of liver disease or liver injury as indicated by an abnormal liver function profile such as SGOT, SGPT, GGT, alkaline phosphate, or serum bilirubin.
* Hepatitis B as indicated by positive HBs Ag or positive anti-HBc IgM result, or Hepatitis C as indicated by positive anti-HCV result.
* History of acute or chronic bronchospastic disease, including asthma and chronic obstructive pulmonary disease, treated or not treated.
* Any surgical or medical condition which might significantly alter the absorption, distribution, or excretion of any drug. The investigator should be guided by evidence of any of the following: History of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding, chronic diarrhoea; History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; History of pancreatic injury or pancreatitis; indications of impaired pancreatic function/injury as indicated by abnormal lipase or amylase; History or presence of impaired renal function as indicated by abnormal creatinine or BUN values or abnormal urinary constituents (e.g., albuminuria); History of urinary obstruction or difficulty in voiding polymorphonuclears <1000/µL or platelets <100'000/µL at inclusion.
* Known history of autoimmune disease such as SLE Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2006-11

PRIMARY OUTCOMES:
Influence of moderate hepatic impairment on the pharmacokinetics of
licarbazepine after single oral administration of 1000 mg licarbazepine (given as 2 x 500
mg IR tablets) in healthy subjects and in moderate hepatic impaired subjects

SECONDARY OUTCOMES:
Influence of moderate hepatic impairment on the pharmacokinetics of the two enantiomers of licarbazepine and the glucuronide conjugates of licarbazepine and its
two enantiomers after single oral administration of 1000 mg licarbazepine (given as 2 x
500 mg IR tablets) in healthy subjects and in moderate hepatic impaired subjects
Safety and tolerability of single oral doses of 1000 mg licarbazepine (given
as 2 x 500 mg IR tablets) in healthy subjects and in moderate hepatic impaired subjects

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Prague, Czechia